CLINICAL TRIAL: NCT00628082
Title: Energetic Abnormalities in Heart Failure With Preserved Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other); British Heart Foundation (Other)
Responsible Party: Prof Michael Frenneaux, University of Birmingham
Other Study IDs: RRK 2996
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Heart Failure, Diastolic
Keywords: Cardiac Energetics; Dynamic Diastolic filling Assessment; Heart Failure with Preserved Ejection Fraction; Arterial and Ventricular Stiffening
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HfpEF: Patients with Heart Failure with preserved ejection fraction
- Control: Healthy Volunteers

SUMMARY:
Up to half of all patients with heart failure are found to have normal pumping function of the heart muscle, but show abnormalities in the way the heart muscle relaxes and fills with blood. These patients often have high blood pressure, and tend to have stiff arteries and stiff heart muscle. We wish to test the hypothesis that these patients have abnormal energy stores in their heart muscle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features consistent with heart failure
* LVEF ≥ 50%, with no evidence of significant valvular disease, no hypertrophic cardiomyopathy, and no evidence of pericardial constriction
* A peak VO2 < 80% predicted, with a pattern of gas exchange on metabolic exercise testing indicating a cardiac cause for limitation

Exclusion Criteria:

* Objective evidence of lung disease on formal lung function testing
* Reversible myocardial ischaemia on contrast-enhanced myocardial stress
* Echocardiography, and evidence of exercise-induced mitral regurgitation
* Obesity (BMI >35) or a locomotor cause for exercise limitation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart Failure Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Complete echocardiographic assessment to assess resting diastolic function | 1 DAY
Assessment of resting large artery function | 1 DAY
Multiple Gated Acquisition Scan | 1 DAY
Cardiac Magnetic Resonance Spectroscopy | 1 DAY
Metabolic Exercise Testing (VO2max) | 1 DAY

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frenneaux, FRCP, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom